CLINICAL TRIAL: NCT05332041
Title: Clinical Assessment of Bioactive Bulk Fill Composite Versus High Viscosity Glass Ionomer Restorations for Restoring Occlusal Carious Lesions of Posterior Teeth in Patients Scheduled for Head and Neck Radiotherapy
Brief Title: Assessment of Bioactive Bulk Fill Composite Versus High Viscosity Glass Ionomer Restorations for Carious Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Neven Ahmed Ebrahim, Neven Ahmed Ebrahim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: USPHS criteria
Record Dates: First submitted 2022-04-06; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Secondary Dental Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Predicta Bioactive bulk fil composite restoration (Experimental): Bioactive bulk fil resin composite dental restoration material
  Interventions: Other: Predicta Bioactive bulk fil composite restoration
- High viscosity glass ionomer (Equia Fil) (Active Comparator): High viscosity dental restoration material
  Interventions: Other: Predicta Bioactive bulk fil composite restoration

INTERVENTIONS:
Other: Predicta Bioactive bulk fil composite restoration — Predicta Bioactive bulk fil resin composite restoration material

SUMMARY:
This trial will be conducted to compare the clinical performance between a new bioactive resin composite material and high viscosity glass ionomer for restoring occlusal carious lesions of posterior teeth in patients scheduled for head and neck radiotherapy.

DETAILED DESCRIPTION:
Inspite of recent developments in the materials' science, some novel materials require direct association with components of the oral cavity for renewal or recharging of the constituents of the restoration to enhance marginal integrity and thus decrease bacterial microleakage, marginal discoloration and postoperative hypersensitivity . There is a constant increase in aesthetic demand for a material that ensures near to perfect adhesion to the tooth surface in order to minimize microleakage and improve marginal integrity. Microleakage forms the basis for predicting the performance of any restorative material Bioactive restorative materials have been introduced for numerous utilizations in dentistry. Among these are fluorides for remineralization; antibacterial resins and restoratives that release and recharge fluorides, phosphate and hydroxyle ions and thus can enhance marginal integrity . Bioactive restorative materials are reported to release more fluoride than glass ionomers. Additionally, they react to pH changes in the mouth by uptaking calcium, phosphate, and fluoride ions to maintain the chemical integrity of the tooth structure.

It is proposed that contemporary bioactive esthetic materials, which associate with oral fluids and show recharge and renewal of restorative material constituents, have the potential to reduce bacterial microleakage and enhance marginal integrity, One possible approach to increase the resistance of restorations to secondary caries formation is to use bioactive materials ( Like predicta bilk fil composite) that contain agents which negatively influence the micro-organisms and/or promote remineralization of tooth structure.

High viscosity glass ionomer (EQUIA Fil) has new technology that contains ultrafine and highly reactive glass diffused within the glass-ionomer fillers to increase and enhance matrix formation. This system allows ion availability and builds a stronger matrix structure with greater physical properties, wear resistance and fluoride release.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion:

1. Patients Scheduled for head and neck radiotherapy.
2. age: ≥18 years.
3. Patients with good likelihood of recall availability.

Tooth inclusion:

1. Permanent premolars or molars.
2. Primary occlusal carious lesions.
3. Vital with positive reaction to cold thermal stimulus.
4. Well-formed and fully-erupted.

Exclusion Criteria:Patient exclusion:

1. Participants with late stage head and neck cancer
2. Concomitant participation in another research study.
3. Inability to comply with study procedures
4. past experience with allergic reactions against any components of the used materials Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.

N 2-Non-vital teeth. 3-Secondary carious lesions

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Secondary caries | one year follow up
  biological outcome